CLINICAL TRIAL: NCT02720575
Title: Evaluation of the Bioavailability of Vitamin D2 in Yeast and Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Michael F. Holick, Professor, Boston University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-833963
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Vitamin D; Bioavailability; Fortified Bread
MeSH Terms: interventions — Bread; Vitamin D

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A (Active Comparator): 50,000 IU of crystalline D2 in 5 capsules.. Vitamin D2 in its natural state consumed orally via capsule
  Interventions: Other: Consumption of capsule/bread with vitamin D
- B (Active Comparator): 50,000 IU of crystalline D3 in 5 capsules.. Vitamin D3 in its natural state consumed orally via capsule
  Interventions: Other: Consumption of capsule/bread with vitamin D
- C (Active Comparator): 50,000 IU of vitamin D2 from vitamin D2 yeast in 5 capsules. Vitamin D generated in yeast. Acts as a comparator to the yeast in bread.
  Interventions: Other: Consumption of capsule/bread with vitamin D
- D (Active Comparator): 50,000 IU of vitamin D2 from yeast cell walls in 5 capsules. Yeast cell walls rich in Vitamin D. Acts as a comparator to the yeast in bread.
  Interventions: Other: Consumption of capsule/bread with vitamin D
- E (Experimental): 50,000 IU of vitamin D2 from 2 slices of bread made from bread. Bread raised with yeast rich in vitamin D. Main experimental arm.
  Interventions: Other: Consumption of capsule/bread with vitamin D
- F (Experimental): 50,000 IU of vitamin D2 from 2 slices of bread. Bread raised with yeast and yeast cell walls rich in vitamin D.
  Interventions: Other: Consumption of capsule/bread with vitamin D

INTERVENTIONS:
Other: Consumption of capsule/bread with vitamin D

SUMMARY:
The objective of this study is to test the bioavailability of vitamin D in bread.

DETAILED DESCRIPTION:
Vitamin D helps in reducing the risk for the development of many chronic diseases. Humans get vitamin D mainly from direct exposure to sunlight, from diet, or from dietary supplements. The bioavailability of vitamin D from dietary supplements has been tested. In one study, subjects had initial vitamin D level of less than 10ng/ml, and it rose to 60ng/ml 24 hours after taking a vitamin D supplement capsule that contained 50,000 IU of vitamin D2. Food contains vitamin D2 or vitamin D3 either naturally or after being fortified. Fortification of dietary products date back to the first half of the 20th century when Steenbock discovered that irradiation of food helped in promoting the healing of rickets in vitamin D deficient rachitic rats. Since that time, companies started to fortify their products to enhance their vitamin D content. In the 1930s Bond Bread fortified its bread with vitamin D2. Recently the FDA approved yeast vitamin D2 which is a yeast that was exposed to ultraviolet radiation. This yeast is active and when used to raise bread the bread contains vitamin D2. The baking process does not affect the vitamin D content. What is unknown is whether the vitamin D2 that is produced in the bread is bioavailable. The purpose of this study is to determine the bioavailability of vitamin D2 that is present in yeast, in bread that was raised with vitamin D2 yeast and vitamin D2 in the cell walls of yeast compared to a vitamin D2 supplement and a vitamin D3 supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adult who are free of any chronic disease
2. Age 18-64 years
3. BMI <30kg/m2
4. No medications or disorders that would affect vitamin D metabolism
5. Women must be on birth control and not pregnant based on negative pregnancy test
6. Ability and willingness to give informed consent and comply with protocol
7. Subjects will be included in the study regardless of their baseline vitamin D level. This is because the level is undetectable unless the subjects is taking high amount of vitamin D, and we will be excluding subjects who are taking pharmacologic doses of vitamin D of >10,000 IUs. Doses of vitamin D in supplements typically contain 400 IUs and up to 1000 IUs. Taking this amount of vitamin D will not significantly raise blood levels of vitamin D from baseline which is usually less than 5 ng/mL. Taking 1000 IUs of vitamin D will raise the blood level by approximately 1-2 ng/mL. Taking a single dose of 50,000 IUs of vitamin D raises the blood level by 50-100 ng/mL. Also a person's vitamin D status i.e. serum 25-hydroxyvitamin D does not affect how vitamin D is absorbed by the intestine nor does it influence the response of oral vitamin D on blood levels of vitamin D which is the goal of this proposal.

Exclusion Criteria:

* 1. Having history of hypercalcemia. 2. Taking over the counter or prescription vitamin D that is greater than 10,000 IUs daily.

  3. Pregnancy. 4. History of intestinal malabsorption. 5. Inability to give informed consent. 6. Chronic hepatic or renal failure. 7. Subjects taking cholestyramine and olestra. 8. Celiac disease. 9. Allergy to wheat or gluten sensitivity.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evidence of serum vitamin D levels proceeding ingestion of bread raised with yeast containing vitamin D | within the fist 24, 48, 72, 96, and 144 hours after ingestion
  The subject blood will be monitored at the above mentioned time frame after consuming vitamin D in capsular or bread form.